CLINICAL TRIAL: NCT00314015
Title: Evaluation of the Success Rate of Immediately Loaded Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/121
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Dental Implants
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with immediately loaded implants. (Experimental)
  Interventions: Procedure: Evaluation of the success rate of implants; Procedure: Questionnaires

INTERVENTIONS:
Procedure: Evaluation of the success rate of implants — Evaluation of the success rate of implants will be followed.
Procedure: Questionnaires — Questionnaires will be used

SUMMARY:
Evaluation of the success rate of immediately loaded implants based on:

* condition of the gingiva
* stability of the implants
* evaluation of the RXs
* questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Patients with immediately loaded implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2008-12-31 (Actual); Study Completion 2008-12-31 (Actual)

PRIMARY OUTCOMES:
Success of implants | Continuous follow-up
Prothetic complications | Continuous follow-up
Opinion of the patient | Continuous follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hugo De Bruyn, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be